CLINICAL TRIAL: NCT00835757
Title: Diffusion Tensor Imaging of Sural Nerves in Diabetic Peripheral Neuropathy"
Brief Title: Diffusion Tensor Imaging of Sural Nerves in Diabetic Peripheral Neuropathy
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Principal Investigator, Rodica Pop-Busui, Associate Professor of Internal Medicine/MEND, University of Michigan
Other Study IDs: 1-2008-1025; JDRF 1-2008-1025
Record Dates: First submitted 2009-02-02; First posted 2009-02-04 (Estimated); Last update posted 2013-12-17 (Estimated); Status verified 2013-12

CONDITIONS: Diabetic Peripheral Neuropathy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Diabetic peripheral neuropathy
- 2: Healthy controls

SUMMARY:
This study aims to validate magnetic resonance imaging and diffusion tensor imaging (MRI/ DTI) analysis as a non-invasive method for the assessment of myelinated nerve fibers loss in diabetic peripheral neuropathy.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of diabetes mellitus diagnosed for more than 6 months as defined by the World Health Organization Classification.
2. Presence of confirmed DPN as defined below.
3. Age between 18-70 years.
4. Have no risk factors for other non-diabetic neuropathies (as determined by medical history, family history, history of medications, occupational history, history of exposure to toxins, physical and neurological examinations).
5. Willingness to provide informed consent and cooperate with the medical procedures for the study.

Inclusion Criteria for Healthy Controls:

1. Age-matched non-obese (BMI < 30) control subjects
2. Normal glucose tolerance
3. Normal blood pressure
4. Normal lipid profile
5. Free of any causes of neuropathy as described above.

Exclusion Criteria:

1. Nursing mothers or pregnant women (excluded by a positive pregnancy test).
2. Patients with a history of previous kidney, pancreas or cardiac transplantation.
3. Patients with a past history of neuropathy (independent of diabetes), or with a disease known to be associated with neuropathy (e.g. end stage renal disease, hepatitis C, systemic lupus erythematosus).
4. Participation in an experimental medication trial within 3 months of starting the study.
5. Subjects with implantable cardioverter defibrillators and other devices that would preclude MRI scanning.
6. Subjects who are unable or unwilling to comply with the experimental protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Two groups of 25 subjects each will be studied: subjects with confirmed diabetic peripheral neuropathy (DPN) and age- and sex-matched healthy controls.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2008-09; Primary Completion 2012-06 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
The difference in means between DTI parameters (FA and MD) measured in the sural nerve between subjects with DPN and healthy control subjects. | 12-18 months

SECONDARY OUTCOMES:
The association between DTI parameters and clinical and electrophysiological measures of DPN | 12-18 months

CONTACTS AND LOCATIONS:
Overall Officials: Rodica Pop-Busui, MD, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States